CLINICAL TRIAL: NCT04454996
Title: Major Achievements in Traditional Chinese Medicine Science and Technology Guidance Projects-Study on the Rule and Mechanism of Treating Functional Gastrointestinal Diseases
Brief Title: Study on the Rule and Mechanism of Treating Functional Gastrointestinal Diseases From the Perspective of Liver and Spleen
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZZ13-ZD-02
Record Dates: First submitted 2020-06-20; First posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Non-erosive Reflux Disease/Diarrheal Irritable Bowel Syndrome
MeSH Terms: conditions — Non-Erosive Reflux Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Non-erosive reflux disease test group (Experimental)
  Interventions: Drug: tong-jiang granules
- Non-erosive reflux disease control group (Placebo Comparator)
  Interventions: Drug: The placebo of tong-jiang granules
- Diarrhea-type irritable bowel syndrome test group (Experimental)
  Interventions: Drug: Chang 'an II Recipe
- Control group with diarrheal irritable bowel syndrome (Placebo Comparator)
  Interventions: Drug: The placebo of Chang 'an II Recipe
- Healthy control group (No Intervention)

INTERVENTIONS:
Drug: tong-jiang granules — This is a kind of compound Chinese medicine granules, 1 bag each time, 3 times a day, treatment for 4 weeks.
  Arms: Non-erosive reflux disease test group
Drug: Chang 'an II Recipe — This is Chang 'an II Prescription granule, 1 bag each time, 3 times a day, treatment for 4 weeks.
  Arms: Diarrhea-type irritable bowel syndrome test group
Drug: The placebo of tong-jiang granules — This is a granule, containing 5% tongyu granule active drug,1 bag each time, 3 times a day, treatment for 4 weeks.
  Arms: Non-erosive reflux disease control group
Drug: The placebo of Chang 'an II Recipe — This is a granule containing 5% chang 'an II,1 bag each time, 3 times a day, treatment for 4 weeks.
  Arms: Control group with diarrheal irritable bowel syndrome

SUMMARY:
To clarify the changes of intestinal flora - gut - brain axis in FGIDs patients represented by NERD disharmony of liver and stomach and IBS-D disharmony of liver and spleen, and confirm that the imbalance between intestinal flora and host co-metabolism is the key to the pathogenesis of functional gastrointestinal disease. To reveal the common mechanism of regulating liver and spleen (stomach) in treating FGIDs dynamic disorder and visceral hypersensitivity by regulating intestinal flora - intestine - brain axis disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers with no abnormal clinical manifestations;
2. Meet the diagnostic criteria of NERD syndrome of disharmony of liver and stomach and IBS-D syndrome of liver depression and spleen deficiency.
3. Aged between 18 and 70.
4. Did not take antibiotics, steroids or other hormones, Chinese herbal preparations (including oral and intravenous administration), microecological preparations or probiotics such as yogurt for nearly a week;
5. Subjects are informed and sign informed consent voluntarily;
6. Have certain reading ability.

Exclusion Criteria:

1. Patients with severe lesions of the heart, liver, kidney and other major organs, hematopoietic system, nervous system or mental diseases;
2. Complicated with other organic diseases of the digestive system (such as peptic ulcer), or systemic diseases that affect the dynamics of the digestive tract (such as hyperthyroidism and diabetes);
3. Ongoing or ongoing use of drugs that may affect gastrointestinal function (antidiarrals, antidepressants, anti-anxiety drugs, intestinal microflora regulation drugs, antibiotics, etc.);
4. Those with a history of allergy to related drugs or severe food allergy used in the research.
5. The body is colonized with metal medical devices. (6) Having a pregnancy plan within three months.

   -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-06-25 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Changes in 7 point Likert scale scores | Baseline, 2 weeks and 4 weeks during treatment period,4 weeks , 8 weeks , 12 weeks and 16 weeks during follow-up period
  The score of patients on the degree of remission of gastroesophageal reflux disease symptoms (acid reflux and heartburn) (1 point for obvious improvement of symptoms, 2 points for improvement of symptoms, 3 points for slight improvement of symptoms, 4 points for no change, 5 points for slight aggravation of symptoms, 6 points for aggravation of symptoms, and 7 points for obvious aggravation of symptoms)
Changes in irritable bowel syndrome symptom severity scale scores | Baseline, 2 weeks and 4 weeks during treatment period,4 weeks , 8 weeks , 12 weeks and 16 weeks during follow-up period
  Irritable bowel syndrome symptom severity scale scores were assessed before and after treatment and during follow-up. The scoring standard is the same as the international standard.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiyuan Hospital of China Academy of Chinese Medical Science, Beijing, Beijing Municipality, China